CLINICAL TRIAL: NCT00350337
Title: Phase II, Randomized, Observer-Blind, Single Center, Controlled Study of Two Doses of Various Formulations of WRAIR Live Attenuated Tetravalent Dengue Vaccine Compared to Placebo Control Administered on 0-6-Month Schedule to Healthy Adults
Brief Title: Safety and Immunogenicity of Various Formulations of Live Attenuated Tetravalent Dengue Vaccine in Healthy US Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WRAIR 1151; GSK 103996 (Other: GalaxoSmithKline); HSRRB A-13291 (Other: USAMRMC HSRRB)
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Pre-transfection F17 (Experimental): 4 monovalent vaccine lots: DEN type 1 45AZ5 PDK-27, Lot 1-1-90 DEN type 2 S16803 PDK-50, Lot 1-1-90 DEN type 3 CH53489 PDK-20 DEN type 4 341750 PDK-6, Lot 1-1-90 in 50% EMEM stabilizer, streptomycin, neomycin and vegetable-derived carbohydrates and amino acids stabilizers for injection.
  Freeze-dried monovalent dengue vaccines were rehydrated with sterile water for injection diluted to match viral concentration of the F17 Post vaccine
  Interventions: Biological: Pre-transfection F17
- Post-transfection F17 (Experimental): 4 monovalent vaccine lots: DEN type 1: 4.9 log10 FFU/mL DEN type 2 : 5.3 log10 FFU/mL DEN type 3: 4.7 log10 FFU/mL DEN type 4: 5.0 log10 FFU/mL in 50% EMEM stabilizer, streptomycin, neomycin and vegetable-derived carbohydrates and amino acids stabilizers for injection.
  Lyophilized, single dose vials and sterile water for injection
  Interventions: Biological: Post-transfection F17
- Post-transfection F19 (Experimental): 4 monovalent vaccine lots: DEN type 1: 4.9 log10 FFU/mL DEN type 2: 5.2 log10 FFU/mL DEN type 3: 4.6 log10 FFU/mL DEN type 4: 4.4 log10 FFU/mL (1:10 dilution) in 50% EMEM-stabilizer, streptomycin, neomycin and vegetable-derived carbohydrates and amino acids stabilizers for injection.
  Lyophilized, single dose vials and sterile water for injection
  Interventions: Biological: Post-transfection F19
- Placebo (Placebo Comparator): A sterile solution of the same EMEM, with phenol red (1:1) and the same virus stabilizer contained in the vaccine. The phenol red dye (phenolsulfonphthalein) is an FDA-accepted vaccine excipient used in vaccines as a pH indicator. The placebo was identical in appearance to the dengue vaccine.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Pre-transfection F17 — Dengue tetravalent Vaccine F17 Pre transfection: 0.5 mL volume per dose, administered at 0 and 6 months via subcutaneous injection
  Arms: Pre-transfection F17
Biological: Post-transfection F17 — Dengue tetravalent Vaccine F17 Post transfection: 0.5 mL volume per dose, administered at 0 and 6 months via subcutaneous injection. For the booster phase of the study, a booster dose was administered at five months to one year following the second dose.
  Arms: Post-transfection F17
Biological: Post-transfection F19 — Dengue tetravalent Vaccine F19 Post transfection: 0.5 mL volume per dose, administered at 0 and 6 months via subcutaneous injection. For the booster phase of the study, a booster dose was administered at five months to one year following the second dose.
  Arms: Post-transfection F19
Other: Placebo — Sterile solution of buffered water (0.9% NaCl), U.S. FDA accepted vaccine excipient, phenol red dye(phenolsulfonphthalein, used in vaccines as a pH indicator); 0.5 mL volume per dose, administered at 0 and 6 months via subcutaneous injection
  Arms: Placebo

SUMMARY:
This descriptive study will evaluate the safety and immunogenicity of 3 different formulations of the WRAIR dengue vaccine compared to a placebo.

DETAILED DESCRIPTION:
Subjects will be randomized into one of 4 groups. One group will receive a placebo vaccine and the others will receive one of 3 different dengue vaccine formations. Each subject will receive two doses six months apart. Study subjects who elect to participate in a mosquito transmissibility component of the study will undergo mosquito feedings during each of the two assigned follow-up visits after vaccine dose 1. All subjects will have 11 venipunctures during 11 visits (i.e., screening plus 10 study visits) over a period of nine months.

A third (booster) dose of post transfection F17 or F19 will be administered approximately 5 to 12 months after dose 2 to all subjects who received one of these formulation for their first two doses. Volunteers will return for a single visit 6 months after receiving their booster dose (long term follow-up)

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female adult 18-45 years at the time of vaccination;
* Free of obvious health problems as established by medical history and physical examination before entering into the study;
* Written informed consent obtained from the subject;
* Able to read the Subject Information Sheet and Consent Form;
* Subjects who the investigator believes can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits) should be enrolled in the study;
* If the subject is female, she must be of non-childbearing potential, i.e. either surgically sterilized or one year post-menopausal; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (i.e. intrauterine contraceptive device; oral contraceptives or other equivalent hormonal contraception, e.g. progestin implantable, cutaneous hormonal patch or injectable contraceptives) for 30 days prior to vaccination, have a negative pregnancy test within 48 hours prior to vaccination and must agree to continue such precautions for 60 days after completion of the vaccination series.

Exclusion Criteria:

* Pregnant or lactating female;
* Female planning to become pregnant or planning to discontinue abstinence or contraceptive precautions;
* History of any neurological or behavioral disorder or seizures, with the exception of a single febrile seizure in childhood;
* History of drug abuse or alcohol consumption (more than 2 drinks per day);
* History of allergic disease/reaction likely to be exacerbated by any component of the vaccine;
* History of urticaria related to mosquito bites requiring medical attention;
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, renal, hematologic or endocrine functional defect, as determined by physical examination or laboratory tests;
* Any confirmed or suspected immunosuppressive or immunodeficient condition;
* Subject seropositive for HBsAg, anti-HCV or anti-HIV;
* Acute disease at the time of enrollment (acute disease is defined as the presence of a moderate or severe illness with or without fever);
* (Vaccine can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e., oral temperature <37.5°C/<99.5°F.)
* Chronic hepatomegaly, right upper quadrant abdominal pain or tenderness;
* Chronic splenomegaly, left upper quadrant abdominal pain or tenderness;
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the study vaccine (includes placebo) or planned use during the study period;
* Planned administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of the study vaccine and ending 30 days after;
* A planned move to a location that will prohibit participating in the trial for 9 months after the initial vaccination;
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 90 days preceding the first dose or planned administration during the study period. For corticosteroids, this will mean prednisone, or equivalent, 0.5 mg/kg/day. Inhaled and topical steroids are allowed;
* Administration of immunoglobulins and/or blood products within 90 days preceding the first dose or planned administration during the study period;
* Any chronic systemic drug therapy to be continued during the study period (except for vitamin/mineral supplements, a single anti-hypertension medication or routine treatment for gastro-esophageal reflux).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2006-04-05 (Actual); Primary Completion 2007-06-20 (Actual); Study Completion 2008-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Thomas, MD, FACP, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

REFERENCES:
- [Derived] Thomas SJ, Eckels KH, Carletti I, De La Barrera R, Dessy F, Fernandez S, Putnak R, Toussaint JF, Sun W, Bauer K, Gibbons RV, Innis BL. A phase II, randomized, safety and immunogenicity study of a re-derived, live-attenuated dengue virus vaccine in healthy adults. Am J Trop Med Hyg. 2013 Jan;88(1):73-88. doi: 10.4269/ajtmh.2012.12-0361. Epub 2012 Dec 3. PMID 23208878

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-transfection F17: 4 monovalent vaccine lots: DEN type 1 45AZ5 PDK-27, Lot 1-1-90 DEN type 2 S16803 PDK-50, Lot 1-1-90 DEN type 3 CH53489 PDK-20 DEN type 4 341750 PDK-6, Lot 1-1-90 in 50% EMEM stabilizer, streptomycin, neomycin and vegetable-derived carbohydrates and amino acids stabilizers for injection.
  Freeze-dried monovalent dengue vaccines were rehydrated with sterile water for injection diluted to match viral concentration of the F17 Post vaccine.
  Pre-transfection F17: Dengue tetravalent Vaccine F17 Pre transfection: 1.0 mL volume per dose, administered at 0 and 6 months via subcutaneous injection.
- Post-transfection F17: DEN type 1: 4.9 log10 FFU/mL DEN type 2 : 5.3 log10 FFU/mL DEN type 3: 4.7 log10 FFU/mL DEN type 4: 5.0 log10 FFU/mL in 50% EMEM stabilizer, streptomycin, neomycin and vegetable-derived carbohydrates and amino acids stabilizers for injection. Lot 1262.
  Lyophilized, single dose vials and sterile water for injection.
  Post-transfection F17: Dengue tetravalent Vaccine F17 Post transfection: 0.5 mL volume per dose, administered at 0 and 6 months via subcutaneous injection. For the booster phase of the study, a booster dose was administered at five months to one year following the second dose.
- Post-transfection F19: DEN type 1: 4.9 log10 FFU/mL DEN type 2: 5.2 log10 FFU/mL DEN type 3: 4.6 log10 FFU/mL DEN type 4: 4.4 log10 FFU/mL (1:10 dilution) in 50% EMEM-stabilizer, streptomycin, neomycin and vegetable-derived carbohydrates and amino acids stabilizers for injection. Tetravalent vaccine lot 1263.
  Lyophilized, single dose vials and sterile water for injection
  Post-transfection F19: Dengue tetravalent Vaccine F19 Post transfection: 0.5 mL volume per dose, administered at 0 and 6 months via subcutaneous injection. For the booster phase of the study, a booster dose was administered at five months to one year following the second dose.
- Placebo: A sterile solution of the same EMEM, with phenol red (1:1) and the same virus stabilizer contained in the vaccine. The phenol red dye (phenolsulfonphthalein) is an FDA-accepted vaccine excipient used in vaccines as a pH indicator. The placebo was identical in appearance to the dengue vaccine. Lot 1249.
  Lyophilized, single dose vials and sterile water for injection.
  Placebo: 0.5 mL volume per dose, administered at 0 and 6 months via subcutaneous injection.
Period: Overall Study
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo
Started | 22 | 22 | 21 | 21
Completed | 17 | 19 | 18 | 21
Not Completed | 5 | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 21 | 21 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 21 | 21 | 86
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (7.75) | 32.8 (6.93) | 33 (8.6) | 35.8 (6.7) | 34.3 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 8 | 10 | 35
  Male | 16 | 11 | 13 | 11 | 51
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 21 | 21 | 86

OUTCOME MEASURES:

1. Primary Outcome: N Antibody, Geometric Mean Titer(GMT) to Dengue Serotypes 1, 2, 3 and 4
Description: GMTs for DEN neut. antibodies -unprimed subjects (primary and booster ATP Cohort for immunogenicity) PRE = Pre dose PI(M1) = Post dose 1, month 1 PII(M7) = Post dose 2, month 7 PRE III = Pre dose 3 PIII(M1) = Post dose 3, month 1
Time Frame: Pre dose 1, 1 month post dose 1, 7 months post dose 2, Pre dose 3 and 1 month post dose 3
Population: Number of subjects with titer within specified range
Measure: Mean (95% Confidence Interval); unit: GMT value
Groups:
- Post-transfection F17: DEN type 1: 4.9 log10 FFU/mL DEN type 2 : 5.3 log10 FFU/mL DEN type 3: 4.7 log10 FFU/mL DEN type 4: 5.0 log10 FFU/mL in 50% EMEM stabilizer, streptomycin, neomycin and vegetable-derived carbohydrates and amino acids stabilizers for injection. Lot 1262.
  Lyophilized, single dose vials and sterile water for injection; 0.5 mL F17Post vaccine
  Post-transfection F17: Dengue tetravalent Vaccine F17 Post transfection: 0.5 mL volume per dose, administered at 0 and 6 months via subcutaneous injection. For the booster phase of the study, a booster dose was administered at five months to one year following the second dose.
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19
Number analyzed (Participants) | 16 | 16 | 15
GMT value
  DEN-1: PRE | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
  DEN-1: PI(M1) | 13 [3 to 53] | 8 [4 to 17] | 55 [11 to 281]
  DEN-1: PII(M7): number analyzed (Participants) | 14 | 15 | 12
  DEN-1: PII(M7) | 195 [57 to 665] | 46 [12 to 175] | 98 [25 to 387]
  DEN-1: PRE III: number analyzed (Participants) | 16 | 6 | 7
  DEN-1: PRE III | NA [NA to NA] — Data not collected for this time point | 10.2 [1.7 to 61.6] | 30.3 [4.6 to 197]
  DEN-1: PIII(M1): number analyzed (Participants) | 16 | 6 | 7
  DEN-1: PIII(M1) | NA [NA to NA] — Data not collected at this time point | 42.7 [8.4 to 217] | 73.3 [19.1 to 280]
  DEN-2: PRE | 2 [2 to 2] | 2 [2 to 2] | 2 [1 to 2]
  DEN-2: P1(M1) | 141 [43 to 460] | 49 [14 to 169] | 168 [41 to 680]
  DEN-2: PII(M7) | 666 [376 to 1179] | 125 [30 to 523] | 226 [70 to 729]
  DEN-2: PRE III | NA [NA to NA] — Data not collected for this time point | 30 [3.9 to 227] | 31.5 [6.3 to 157]
  DEN-2: PIII(M1) | NA [NA to NA] — Data not collected for this time point | 100 [13.3 to 749] | 194.5 [56.1 to 674]
  DEN-3: PRE | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
  DEN-3: PI(M1) | 13 [4 to 38] | 9 [4 to 18] | 16 [5 to 50]
  DEN-3: PII(M7) | 78 [21 to 286] | 27 [8 to 98] | 48 [13 to 177]
  DEN-3: PRE III | NA [NA to NA] — Data not collected for this time point | 4.1 [1.0 to 16.9] | 10.1 [2.5 to 40.9]
  DEN-3: PIII(M1) | NA [NA to NA] — Data not collected for this time point | 28.2 [3.2 to 249.4] | 19.7 [5.6 to 69.8]
  DEN-4: PRE | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
  DEN-4: PI(M1) | 16 [4 to 74] | 30 [6 to 150] | 28 [6 to 128]
  DEN-4: PII(M7) | 271 [53 to 1378] | 62 [14 to 284] | 41 [10 to 176]
  DEN-4: PRE III | NA [NA to NA] — Data not collected for this time point | 17.3 [0.6 to 491.9] | 12.1 [1.0 to 1466.2]
  DEN-4: PIII(M1) | NA [NA to NA] — Data not collected for this time point | 44.4 [3.7 to 539.2] | 32.2 [4.5 to 232.2]

2. Primary Outcome: Percentage of Subjects Seropositive for Dengue Serotypes 1, 2, 3 and 4
Description: Serpositivity rates for DEN neut. antibodies -unprimed subjects (primary and booster ATP Cohort for immunogenicity) PRE = Pre dose PI(M1) = Post dose 1, month 1 PII(M7) = Post dose 2, month 7 PRE III = Pre dose 3 PIII(M1) = Post dose 3, month 1
Time Frame: Pre dose 1, 1 month post dose 1, 7 months post dose 2, Pre dose 3 and 1 month post dose 3
Population: Vaccinated subjects for whom assay results were available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19
Number analyzed (Participants) | 16 | 16 | 15
percentage of participants
  DEN-1: PRE | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  DEN-1: PI(M1) | 43.8 [19.8 to 70.1] | 37.5 [15.2 to 64.6] | 66.7 [38.4 to 88.2]
  DEN-1: PII(M7) | 92.9 [66.1 to 99.8] | 73.3 [44.9 to 92.2] | 83.3 [51.6 to 97.9]
  DEN-1: PRE III | NA [NA to NA] — Data not collected for this time point | 66.7 [22.3 to 95.7] | 71.4 [29.0 to 96.3]
  DEN-1: PIII(M1) | NA [NA to NA] — Data not collected for this time point | 83.3 [35.9 to 99.6] | 100 [59.0 to 100]
  DEN-2: PRE | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  DEN-2: PI(M1) | 87.5 [61.7 to 98.4] | 68.8 [41.3 to 89.0] | 86.7 [59.5 to 98.3]
  DEN-2: PII(M7) | 100 [76.8 to 100] | 80.0 [51.9 to 95.7] | 100 [73.5 to 100]
  DEN-2: PRE III | NA [NA to NA] — Data not collected for this time point | 66.7 [22.3 to 95.7] | 57.1 [18.4 to 90.1]
  DEN-2: PIII(M1) | NA [NA to NA] — Data not collected for this time point | 83.3 [35.9 to 99.6] | 100 [59.0 to 100]
  DEN-3: PRE | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  DEN-3: PI(M1) | 50.0 [24.7 to 75.3] | 50.0 [24.7 to 75.3] | 60.0 [32.3 to 83.7]
  DEN-3: PII(M7) | 71.4 [41.9 to 91.6] | 66.7 [38.4 to 88.2] | 83.3 [51.6 to 97.9]
  DEN-3: PRE III | NA [NA to NA] — Data not collected for this time point | 16.7 [0.4 to 64.1] | 42.9 [9.9 to 81.6]
  DEN-3: PIII(M1) | NA [NA to NA] — Data not collected for this time point | 83.3 [35.9 to 99.6] | 57.1 [18.4 to 90.1]
  DEN-4: PRE | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  DEN-4: PI(M1) | 37.5 [15.2 to 64.6] | 56.3 [29.9 to 80.2] | 53.3 [26.6 to 78.7]
  DEN-4: PII(M7) | 78.6 [49.2 to 95.3] | 73.3 [44.9 to 92.2] | 66.7 [34.9 to 90.1]
  DEN-4: PRE III | NA [NA to NA] — Data not collected for this time point | 33.3 [4.3 to 77.7] | 42.9 [9.9 to 81.6]
  DEN-4: PIII(M1) | NA [NA to NA] — Data not collected for this time point | 83.3 [35.9 to 99.6] | 57.1 [18.4 to 90.1]

3. Primary Outcome: Occurrence of Any, and Grade 3 Solicited Adverse Events (AEs) Within 21 Days Follow-up After Dose 1 of Study Vaccine
Description: Diary cards, digital thermometers, and small rulers were provided to subjects to record local and general solicited symptoms(pain, redness and swelling at the injection site, fatigue, headache, pain behind the eyes, abdominal pain, nausea, vomiting, muscle aches, joint aches, rash, photophobia and pruritis) and oral temperature taken daily for 21 days (days 0 through 20). The observations were to be recorded each evening and account for the previous 24 hours. If multiple temperature measurements were taken throughout the day, the maximum temperature was to be recorded.
Time Frame: 21 days following 1st vaccination dose
Measure: Number; unit: participants
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo
Number analyzed (Participants) | 22 | 22 | 21 | 21
participants
  Any Grade 3 symptoms | 1 | 1 | 4 | 3
  General Grade 3 symptoms | 0 | 0 | 3 | 2
  Local Grade 3 symptoms | 1 | 1 | 1 | 2

4. Secondary Outcome: Occurrence of Any, and Grade 3 Solicited Adverse Events (AEs) Within 21 Days Follow-up After Dose 2 of Study Vaccine;
Time Frame: within 21 days after vaccination
Population: Subjects with sufficient data to perform safety analysis
Measure: Number; unit: participants
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo
Number analyzed (Participants) | 16 | 19 | 18 | 20
participants
  Any Grade 3 symptoms | 1 | 1 | 1 | 0
  General Grade 3 symptoms | 1 | 1 | 1 | 0
  Local Grade 3 symptoms | 0 | 0 | 0 | 0

5. Secondary Outcome: Unsolicited Adverse Events Within 31 Days After Each Dose of Study Vaccine Dose
Description: Summary of Unsolicited Adverse Events within 31 days after each dose of study vaccine dose (Primary total vaccinated cohort)
Time Frame: within 31 days of study vaccine
Measure: Number; unit: Number of AEs
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo
Number analyzed (Participants) | 22 | 22 | 21 | 21
Number of AEs
  Any symptoms classified by MedDRA | 27 | 17 | 24 | 30
  Any symptoms reported | 27 | 17 | 24 | 31
  Grade 3 symptoms classified by MedDRA | 1 | 2 | 3 | 2
  Grade 3 symptoms reported | 1 | 2 | 3 | 2
  Casually related symptoms classified by MedDRA | 6 | 1 | 3 | 6
  Casually related symptoms reported | 6 | 1 | 3 | 7
  Grade 3 and casually related symptoms reported | 0 | 0 | 0 | 1

6. Secondary Outcome: Occurrence of Serious Adverse Events (SAEs) Throughout the Entire Study Period.
Description: Serious adverse events will be recorded throughout the entire study period. Subjects instructed to contact the investigator immediately should they manifest any signs or symptoms they perceive as serious. An identification card and a set of phone numbers to contact study staff 24 hours a day, 7 days a week given to subjects.
Time Frame: Days 0 to 270
Measure: Number; unit: participants
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo
Number analyzed (Participants) | 22 | 22 | 21 | 21
participants | 0 | 2 | 1 | 1

7. Secondary Outcome: Occurrence of Abnormal Findings at Physical Examination After Each Vaccine Dose
Description: Abnormal findings at DEN physical examination were defined as:
  rash, generalized rash, hemorrhages (skin, conjunctival or mucosal), conjunctival injection, hepatomegaly, splenomegaly or lymphadenopathy; generalized lymphadenopathy (palpable lymph nodes in 4 or more of the following locations: cervical, axillary, inguinal or other with right and left sides considered as separate locations) positive tourniquet test (WHO criterion of 20 or more petechiae per 2.5 cm square)Results were reported positive/negative using the WHO criterion.
Time Frame: throughout the 202 day study
Measure: Number; unit: participants
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo
Number analyzed (Participants) | 22 | 22 | 21 | 21
participants
  Rash | 3 | 1 | 3 | 0
  Generalized Rash | 1 | 0 | 2 | 0
  Skin Hemorrhage | 0 | 0 | 0 | 1
  Conj. Hemorrhage | 0 | 0 | 0 | 1
  Conj. Injection 2 | 2 | 1 | 2 | 1
  Mucosal Hemorrhage | 2 | 1 | 1 | 1
  Lymphadenopathy | 4 | 6 | 7 | 4
  Generalized Lymphadenopathy | 0 | 1 | 0 | 1
  Hepatomegaly | 2 | 3 | 6 | 4
  Splemonegaly | 0 | 1 | 1 | 2

8. Secondary Outcome: Percentage of Subjects With Suspected and Confirmed Dengue Reported During the 31-day Post-vaccination Period (Total Vaccinated Cohort)
Description: The case definition of confirmed dengue used in this protocol requires fever (equivalent to an oral temperature ≥38.0ºC/≥ 100.4ºF) for three or more successive days, at least two of the signs or symptoms consistent with "suspected dengue" occurring during the period of fever, at least one clinical laboratory abnormality, and DEN viremia detected by RTqPCR. Cases not meeting all criteria were not considered "confirmed dengue." The percentage of subjects with suspected or confirmed dengue were tabulated by group after each vaccination.
Time Frame: Days 0-30 post vaccination periods (total vaccinated cohort)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo
Number analyzed (Participants) | 22 | 22 | 21 | 21
percentage of participants
  Dose 1: Suspected Dengue | 4.5 [0.1 to 22.8] | 0 [0.0 to 15.4] | 0 [0.0 to 16.1] | 4.8 [0.1 to 23.8]
  Dose 1: Confirmed Dengue | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 16.1] | 0 [0.0 to 16.1]
  Dose 2: Suspected Dengue | 0 [0.0 to 19.5] | 0 [0.0 to 17.6] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]
  Dose 2: Confirmed Dengue | 0 [0.0 to 19.5] | 0 [0.0 to 17.6] | 0 [0.0 to 18.5] | 0 [0.0 to 16.8]

9. Secondary Outcome: Neutralizing Antibody Sero-response to Each Dengue Serotype After Each Dose
Description: Sero-response defined as:
  For initially seronegative(S-) subjects, antibody titer >=10 DE50 at PI(M1) For initially seropositive(S+) subjects, antibody titer at PI(M1) >=4 fold the pre-vacciniation neut. antibody titer
Time Frame: Days 0 to 270
Population: Vaccinated subjects for whom assay results were available.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo
Number analyzed (Participants) | 16 | 20 | 18 | 19
percentage of responders
  S- (prior to vaccination) DEN-1 Month 1 | 43.8 [19.8 to 70.1] | 35.3 [14.2 to 61.7] | 66.7 [38.4 to 88.2] | 0 [0.0 to 18.5]
  S+(prior to vaccination) DEN-1 Month 1 | 75 [19.4 to 99.4] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 97.5]
  S- (prior to vaccination) DEN-2 Month 1 | 87.5 [61.7 to 98.4] | 70.6 [44.0 to 89.7] | 86.7 [59.5 to 98.3] | 0 [0.0 to 20.6]
  S+ (prior to vaccination) DEN-2 Month 1 | 50 [6.8 to 93.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0 [0.0 to 70.8]
  S- (prior to vaccination) DEN-3 Month 1 | 50.0 [24.7 to 75.3] | 50.0 [24.7 to 75.3] | 60.0 [32.3 to 83.7] | 0 [0.0 to 18.5]
  S+ (prior to vaccination) DEN-3 Month 1 | 75 [19.4 to 99.4] | 0 [0.0 to 60.2] | 33.3 [0.8 to 90.6] | 0 [0.0 to 97.5]
  S- (prior to vaccination) DEN-4 Month 1 | 37.5 [15.2 to 64.6] | 52.9 [27.8 to 77.0] | 53.3 [26.3 to 78.7] | 11.1 [1.4 to 34.7]
  S- (prior to vaccination) DEN-5 Month 1 | 75.0 [19.4 to 99.4] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0 [0.0 to 97.5]

10. Secondary Outcome: Neutralizing Antibody Sero-response to Each Dengue Serotype After Each Dose (Continued)
Description: as for outcome 9
Time Frame: Days 0 to 270
Population: Vaccinated subjects for whom assay results were available.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo
Number analyzed (Participants) | 16 | 18 | 15 | 19
percentage of responders
  S- (prior to vaccination) DEN-1 Month 7 | 92.9 [66.1 to 99.8] | 73.3 [44.9 to 92.2] | 83.3 [51.6 to 97.9] | 5.6 [0.1 to 27.3]
  S+(prior to vaccination) DEN-1 Month 7 | 50.0 [1.3 to 98.7] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 97.5]
  S- (prior to vaccination) DEN-2 Month 7 | 100 [76.8 to 100] | 80.0 [51.9 to 95.7] | 100 [73.5 to 100] | 0 [0.0 to 20.6]
  S+ (prior to vaccination) DEN-2 Month 7 | 0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0 [0.0 to 70.8]
  S- (prior to vaccination) DEN-3 Month 7 | 71.4 [41.9 to 91.6] | 66.7 [38.4 to 88.2] | 83.3 [51.6 to 97.9] | 5.6 [0.1 to 27.3]
  S+ (prior to vaccination) DEN-3 Month 7 | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0 [0.0 to 97.5]
  S- (prior to vaccination) DEN-4 Month 7 | 78.6 [49.2 to 95.3] | 73.3 [44.9 to 92.2] | 66.7 [34.9 to 90.1] | 0 [0.0 to 18.5]
  S- (prior to vaccination) DEN-5 Month 7 | 50.0 [1.3 to 98.7] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 0 [0.0 to 97.5]

11. Secondary Outcome: Occurrence of Measurable Dengue Viremia at Specified Time Points Following Each Vaccine Dose.
Description: For vireimia:
  Negative = GEQ/µl result is equal to zero Undetermined = GEQ/µL result is below LOD Positive = GEQ/µL result is >= LOD
Time Frame: Days 0 to 270
Measure: Number; unit: participants
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo
Number analyzed (Participants) | 22 | 22 | 21 | 21
participants
  DEN-1 Dose 1 - Positive | 0 | 0 | 0 | 0
  DEN-1 Dose 1 - Undetermined | 2 | 1 | 2 | 1
  DEN-1 Dose 1 - Negative | 18 | 21 | 19 | 20
  DEN-1 Dose 1 - Missing | 2 | 0 | 0 | 0
  DEN-1 Dose 2 - Positive | 0 | 0 | 0 | 0
  DEN-1 Dose 2 - Undetermined | 1 | 2 | 2 | 1
  DEN-1 Dose 2 - Negative | 15 | 17 | 16 | 19
  DEN-1 Dose 2 - Missing | 6 | 3 | 3 | 1
  DEN-1 Overall Subject - Positive | 0 | 0 | 0 | 0
  DEN-1 Overall Subject - Undetermined | 3 | 3 | 3 | 2
  DEN-1 Overall Subject - Negative | 13 | 16 | 15 | 18
  DEN-1 Overall Subject - Missing | 6 | 3 | 3 | 1
  DEN- 2 Dose 1 - Positive | 0 | 0 | 0 | 0
  DEN- 2 Dose 1 - Undetermined | 1 | 1 | 0 | 0
  DEN- 2 Dose 1 - Negative | 18 | 20 | 19 | 19
  DEN- 2 Dose 1 - Missing | 3 | 1 | 2 | 2
  DEN- 2 Dose 2 - Positive | 0 | 0 | 0 | 0
  DEN- 2 Dose 2 - Undetermined | 0 | 1 | 1 | 0
  DEN- 2 Dose 2 - Negative | 15 | 17 | 15 | 18
  DEN- 2 Dose 2 - Missing | 7 | 4 | 5 | 3
  DEN- 2 Overall Subject - Positive | 0 | 0 | 0 | 0
  DEN- 2 Overall Subject - Undetermined | 0 | 2 | 1 | 0
  DEN- 2 Overall Subject - Negative | 15 | 16 | 15 | 18
  DEN- 2 Overall Subject - Missing | 7 | 4 | 5 | 3
  DEN- 3 Dose 1 - Postive | 0 | 0 | 0 | 0
  DEN- 3 Dose 1 - Undetermine | 0 | 0 | 0 | 0
  DEN- 3 Dose 1 - Negative | 20 | 22 | 21 | 21
  DEN- 3 Dose 1 - Missing | 2 | 0 | 0 | 0
  DEN- 3 Dose 2 - Postive | 0 | 0 | 0 | 0
  DEN- 3 Dose 2 - Undetermine | 0 | 0 | 0 | 0
  DEN- 3 Dose 2 - Negative | 16 | 19 | 18 | 20
  DEN- 3 Dose 2 - Missing | 6 | 3 | 3 | 1
  DEN- 3 Overall Subject - Positive | 0 | 0 | 0 | 0
  DEN- 3 Overall Subject - Undetermined | 0 | 0 | 0 | 0
  DEN- 3 Overall Subject - Negative | 16 | 19 | 18 | 20
  DEN- 3 Overall Subject - Missing | 6 | 3 | 3 | 1
  DEN- 4 Dose 1 - Positive | 2 | 1 | 0 | 0
  DEN- 4 Dose 1 - Undetermined | 1 | 1 | 1 | 0
  DEN- 4 Dose 1 - Negative | 17 | 20 | 20 | 21
  DEN- 4 Dose 1 - Missing | 2 | 0 | 0 | 0
  DEN- 4 Dose 2 - Postive | 3 | 0 | 0 | 0
  DEN- 4 Dose 2 - Undetermined | 0 | 0 | 0 | 0
  DEN- 4 Dose 2 - Negative | 13 | 19 | 18 | 20
  DEN- 4 Dose 2 - Missing | 6 | 3 | 3 | 1
  DEN- 4 Overall Subject - Positive | 5 | 1 | 0 | 0
  DEN- 4 Overall Subject - Undetermined | 1 | 1 | 1 | 0
  DEN- 4 Overall Subject - Negative | 11 | 111 | 17 | 20
  DEN- 4 Overall Subject - Missing | 5 | 3 | 3 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms were assessed within the 21 day follow-up period (primary and booster total vaccinated cohort). Unsolicited symptoms were assessed within the 31 day post vaccination period (total vaccinated cohort).
Groups:
- Post-transfection F17: monovalent vaccine lots: DEN type 1: 4.9 log10 FFU/mL DEN type 2 : 5.3 log10 FFU/mL DEN type 3: 4.7 log10 FFU/mL DEN type 4: 5.0 log10 FFU/mL in 50% EMEM stabilizer, streptomycin, neomycin and vegetable-derived carbohydrates and amino acids stabilizers for injection.
  Lyophilized, single dose vials and sterile water for injection
- Post-transfection F19: 4 monovalent vaccine lots: DEN type 1: 4.9 log10 FFU/mL DEN type 2: 5.2 log10 FFU/mL DEN type 3: 4.6 log10 FFU/mL DEN type 4: 4.4 log10 FFU/mL (1:10 dilution) in 50% EMEM-stabilizer, streptomycin, neomycin and vegetable-derived carbohydrates and amino acids stabilizers for injection.
  Lyophilized, single dose vials and sterile water for injection; 0.5 mL F19 vaccines
- Placebo: A sterile solution of the same EMEM, with phenol red (1:1) and the same virus stabilizer contained in the vaccine. The phenol red dye (phenolsulfonphthalein) is an FDA-accepted vaccine excipient used in vaccines as a pH indicator. The placebo was identical in appearance to the dengue vaccine.
  0.5 mL for placebo
Arm/Group | Pre-transfection F17 | Post-transfection F17 | Post-transfection F19 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 2/22 | 1/21 | 1/21
Other Adverse Events (participants affected / at risk) | 19/22 | 19/22 | 16/21 | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-transfection F17 (N=22) | Post-transfection F17 (N=22) | Post-transfection F19 (N=21) | Placebo (N=21)
axonal demyelinating polyneuropathy/bilateral upper and lower extremeties (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rule out cerebral bleed secondary to assualt trauma (physical assault) (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-transfection F17 (N=22) | Post-transfection F17 (N=22) | Post-transfection F19 (N=21) | Placebo (N=21)
Pain (General disorders) | 9 (9) | 3 (3) | 5 (5) | 5 (5)
Redness (Injury, poisoning and procedural complications) | 8 (8) | 3 (3) | 5 (5) | 5 (5)
Swelling (Injury, poisoning and procedural complications) | 7 (7) | 4 (4) | 5 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (5) | 5 (5) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) | 3 (3) | 3 (3)
Fatigue (General disorders) | 10 (10) | 9 (9) | 6 (6) | 7 (7)
Fever >37.5ºC (General disorders) | 5 (5) | 7 (7) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 14 (14) | 11 (11) | 10 (10) | 9 (9)
Muscle aches (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (6) | 5 (5) | 4 (4) | 2 (2)
Pain behind the eyes (Eye disorders) | 4 (4) | 7 (7) | 5 (5) | 3 (3)
Photophobia (Eye disorders) | 4 (4) | 3 (3) | 5 (5) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 3 (3) | 3 (3) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth ache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site hemorrage (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (14) | 0 (0) | 0 (0) | 0 (0)
Fungal rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ejaculation failure (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin warm (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Physical assault (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes